CLINICAL TRIAL: NCT02969382
Title: A 4-Week, Randomized, Double-blind, Parallel-group, Placebo-controlled, Flexibly-dosed, Multicenter Study to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Adult Subjects With Schizophrenia
Brief Title: A Study to Evaluate the Efficacy and Safety of SEP-363856 in Acutely Psychotic Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP361-201; 2016-001555-41 (EudraCT Number)
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Results first posted 2021-09-22 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — SEP-363856

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SEP-363856 (Experimental): SEP-363856 capsule (50 mg or 75 mg) once daily
  Interventions: Drug: SEP-363856
- Placebo (Placebo Comparator): Placebo capsule once daily
  Interventions: Drug: Placebo - Cap

INTERVENTIONS:
Drug: SEP-363856 — One SEP-363856 capsule (50 mg or 75 mg) daily for four weeks
  Arms: SEP-363856
Drug: Placebo - Cap — One Placebo capsule daily for 4 weeks
  Arms: Placebo

SUMMARY:
A study to evaluate the efficacy and safety of an experimental drug (SEP-363856) in acutely psychotic adults with schizophrenia

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, parallel-group, flexibly-dosed, study evaluating the efficacy and safety of SEP-363856 in acutely psychotic adult subjects with schizophrenia using SEP-363856 (50 or 75 mg/day [ie, once daily]) versus placebo over a 4-week treatment period. Primary hypoathesis to be tested: H0: μSEP = μPBO versus H1: μSEP ≠ μPBO, where μSEP and μPBO are the mean changes from Baseline at Week 4 in PANSS total score for the SEP-363856 and placebo arms, respectively. Subjects who complete study SEP361-201 may be eligible to enroll in the open-label extension study SEP361-202.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must give written informed consent and privacy authorization prior to participation in the study. Separate consent will be obtained from a caregiver or legal guardian if required by local law.
2. Subject must be willing and able to comply with the study procedures and visit schedules, including required hospitalization for the washout period and the double-blind treatment period, and must be able to understand and follow verbal and written instructions.
3. Male or female subject between 18 to 40 years of age (inclusive) at the time of consent.
4. Subject meets DSM-5 criteria for schizophrenia as established by clinical interview (using the DSM-5 as a reference and confirmed using the SCID-CT). The duration of the subject's illness whether treated or untreated must be ≥ 6 months.
5. Subject must have a CGI-S score ≥ 4 (moderate or greater) at screening and Baseline (Day 1).
6. Subject must have a PANSS total score ≥ 80 and a PANSS item score ≥ 4 (moderate) on 2 or more of the following PANSS items: delusions, conceptual disorganization, hallucinations, and unusual thought content at screening and Baseline (Day 1).
7. Subject has an acute exacerbation of psychotic symptoms (no longer than 2 months).

   • Subject has marked deterioration of functioning in one or more areas, such as occupational, social, or personal care or hygiene.

   • Subject requires hospitalization for an acute psychotic exacerbation at the time of screening or has been hospitalized for the purpose of treating an acute psychotic exacerbation for no more than 2 consecutive weeks immediately before screening.

   Subjects who have been hospitalized for more than 2 weeks for reasons unrelated to an acute psychotic exacerbation may be included if such a hospitalization was for a condition other than an acute psychotic relapse. For example, subjects in a long-term hospital setting who have an acute exacerbation and are transferred to an acute unit are eligible for the study.
8. Subject has had no more than 2 prior hospitalizations for the treatment of an acute exacerbation of schizophrenia (not including the current hospitalization) This history must be confirmed based on report by a reliable informant (eg., caregiver or family member) or medical records available at the time of screening.
9. Subject's BMI must be at least 18 kg/m2 but no more than 35 kg/m2.
10. Female subject must have a negative serum pregnancy test at screening.11. Female subject of reproductive potential agrees to remain abstinent or use adequate and reliable contraception throughout the study and for at least 30 days after the last dose of study drug has been taken. In the Investigator's judgment, the subject will adhere to this requirement.

    1. Adequate contraception is defined as continuous use of either two barrier methods (eg, condom and spermicide or diaphragm with spermicide) or a hormonal contraceptive.

       Acceptable hormonal contraceptives include the following: a) contraceptive implant (such as Norplant®) implanted at least 90 days prior to screening; b) injectable contraception (such as medroxyprogesterone acetate injection) given at least 14 days prior to screening; or c) oral contraception taken as directed for at least 30 days prior to screening.
    2. Subjects who are of non-reproductive potential, ie, subject who is surgically sterile, has undergone tubal ligation, or is postmenopausal (defined as at least 12 months of spontaneous amenorrhea or between 6 and 12 months of spontaneous amenorrhea with follicle stimulating hormone (FSH) concentrations within postmenopausal range as determined by laboratory analysis) are not required to remain abstinent or use adequate contraception.
11. Female subject of reproductive potential agrees to remain abstinent or use highly effective and reliable contraception throughout the study and for at least 30 days after the last dose of study drug has been taken (See Section 21 Appendix II Highly Effective Protocol SEP361-201, Version 3.01 SEP-363856 Confidential and Proprietary 36 17 August 2017 Contraceptive procedures). In the Investigator's judgment, the subject will adhere to this requirement.
12. Male subjects with female partner(s) of childbearing potential must agree to avoid fathering a child and use highly effective methods of birth control (outlined in Section 21) from screening until at least 30 days after the last study drug administration.
13. Subject must be able and agree to remain off prior antipsychotic medication for the duration of the study.
14. Subject must have a total score < 5 on the SAS at Baseline (Day 1).
15. Subject is, in the opinion of the Investigator, generally healthy based on screening medical history, PE, neurological examination, vital signs, clinical laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, thyroid panel, and serum prolactin).
16. Subject has had a stable living arrangement at the time of screening and agrees to return to a similar living arrangement after discharge. This criterion is not meant to exclude subjects who have temporarily left a stable living arrangement (eg, due to psychosis). Such subjects remain eligible to participate in this protocol. Chronically homeless subjects should not be enrolled.
17. Subject must agree to comply with all restrictions for the required length of time

Exclusion Criteria:

1. Subject answers "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at or during the Screening period (ie, in the past one month) and/or at Baseline (ie, since last visit).

2. Subject does not tolerate venipuncture or has poor venous access that would cause difficulty for collecting blood samples.

3. Subject is currently participating, or has participated in, a study with an investigational or marketed compound or device within 6 months prior to signing the informed consent, or has participated in 2 or more studies within 24 months prior to signing informed consent.

4. Subject has previously received SEP-363856. 5. Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in the study:

1. Hematological (including deep vein thrombosis) or bleeding disorder, renal, metabolic, endocrine, pulmonary, gastrointestinal, urological, cardiovascular, hepatic, neurologic, or allergic disease that is clinically significant or unstable (except for untreated, asymptomatic, seasonal allergies at time of dosing).
2. Subject has a history of neuroleptic malignant syndrome. Protocol SEP361-201, Version 3.01 SEP-363856 Confidential and Proprietary 37 17 August 2017
3. Subject has a history of malignancy within 5 years prior to the Screening visit, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Pituitary tumors of any duration are excluded.
4. Disorder or history of a condition, or previous gastrointestinal surgery (eg, cholecystectomy, vagotomy, bowel resection, or any surgical procedure) that may interfere with drug absorption, distribution, metabolism, excretion, gastrointestinal motility, or pH, or a clinically significant abnormality of the hepatic or renal system, or a history of malabsorption.
5. Subject has Alcohol or Substance Abuse Disorder (DSM-5 criteria). The only exceptions include caffeine or nicotine.
6. Subject has a clinically significant abnormal 12-lead ECG that may jeopardize the subject's ability to complete the study or a screening 12-lead ECG demonstrating any one of the following: heart rate > 100 beats per minute, QRS > 120 ms, QT interval corrected for heart rate using Fridericia's formula (QTcF) > 450 ms (males), QTcF > 470 ms (females), or PR > 220 ms.
7. Subjects with known history of human immunodeficiency virus (HIV) seropositivity.6. 6. Female subject who is pregnant or lactating.

   7. Subject who has a lifelong history or presence of symptoms consistent with a major psychiatric disorder other than schizophrenia as defined by DSM-5. Exclusionary disorders include but are not limited to alcohol use disorder (within past 12 months), substance (other than nicotine or caffeine) use disorder within past 12 months, major depressive disorder, bipolar depression, mania, schizoaffective disorder, obsessive compulsive disorder, posttraumatic stress disorder. Previous or current symptoms of mild to moderate mood dysphoria or anxiety are allowed so long as these symptoms have not been a focus of primary treatment.

   8. Subject tests positive for drugs of abuse at screening, however, a positive test for amphetamines, barbiturates, opiates, benzodiazepines may not result in exclusion of subjects if the investigator determines that the positive test is as a result of prescription medicine(s). In the event a subject tests positive for cannabinoids (tetrahydrocannabinol), the Investigator will evaluate the subject's ability to abstain from using this substance during the study. This information will be discussed with the Medical Monitor prior to study enrollment.

   9. Subject is at significant risk of harming self, others or objects based on the Investigator's judgment.

   10. Subject has attempted suicide within 3 months prior to screening. 11. Subject is involuntarily hospitalized. 12. Subject has received depot antipsychotics unless the last injection was at least one treatment cycle or at least 30 days (whichever is longer), prior to the screening phase.

   13. Subject is judged to be resistant to antipsychotic treatment by the Investigator, based on failure to respond to 2 or more marketed antipsychotic agents, given at adequate dose for at least 4 weeks within a 1 year period prior to Screening.

   14. Subject has a history of treatment with clozapine for refractory psychosis and/or subject has been treated with clozapine (for any reason) within 4 months of Screening.

   15. Subject is receiving a total dose of antipsychotic medication equivalent to > 12.0 mg/day of haloperidol at Screening (see Section 22, Appendix III for table of haloperidol dose equivalents). Subject may be eligible if such treatment is less than 2 weeks in duration after consultation with the Medical Monitor.

   16. Subject has received electroconvulsive therapy treatment within the 3 months prior to screening or is expected to require ECT during the study.

   17. Subject takes or has taken other disallowed recent or concomitant medications (see Section 10.3). Subjects must taper off antipsychotic medications by Day -1.

   18. Subject has a history of allergic reaction or suspected sensitivity to any substance that is contained in the formulation (gelatin).

   19. Subject has any clinically significant abnormal laboratory values (hematology, serum chemistry, urinalysis, lipid panel, coagulation panel, thyroid panel, and serum prolactin (Note: abnormal findings that may be clinically significant or of questionable significance will be discussed with the Medical Monitor prior to including subject).

   20. Subject demonstrates evidence of acute hepatitis, clinically significant chronic hepatitis, or evidence of clinically significant impaired hepatic function through clinical and laboratory evaluation.

   Note: Subjects with serum alanine transaminase (ALT) or aspartate transaminase (AST) levels ≥ 3 times the upper limit of the reference ranges provided by the central laboratory require retesting. If on retesting, the laboratory value remains ≥ 3 times the upper limit, the subject will be excluded.

   21. Subject has a serum blood urea nitrogen (BUN) or serum creatinine (Cr) value ≥ 1.5 times the upper limit of normal for the reference range.

   22. Subject has experienced significant blood loss (≥ 473 mL) or donated blood within 60 days prior to first dose of study drug; has donated plasma within 72 hours prior to the first dose of study drug or intends to donate plasma or blood or undergo elective surgery during study participation or within 60 days after the last study visit.

   23. Subject has used disallowed prescription or disallowed nonprescription drugs, vitamins, or dietary or herbal supplements within 14 days prior to dosing or anticipates the need for any disallowed medication during their participation in this study [exception: female subjects who are taking oral, patch, or intrauterine device (IUD) hormonal contraceptives, or progestin implant or injection].

   24. Subject is a staff member or the relative of a staff member. 25. Subjects with a fasting blood glucose at screening ≥ 126 mg/dL (7.0 mmol/L) or HbA1c ≥ 6.5% will be excluded.

   26. Subject has a prolactin concentration > 100 ng/mL at screening or has a history of pituitary adenoma. NOTE: Subjects with prolactin levels > 100 ng/mL and ≤ 200 ng/mL Protocol SEP361-201, Version 3.01 SEP-363856 Confidential and Proprietary 39 17 August 2017 at the Screening visit are permitted to enroll after discussion with the Medical Monitor to ensure exclusion of non-psychotropic drug-related causes of elevated prolactin levels.

   27. .Subject is in the opinion of the Investigator, unsuitable in any other way to participate in this study.

   Randomization Criteria
   1. Subject must have a PANSS total score ≥ 80 at Baseline (Day 1).
   2. Subject must have a PANSS item score ≥ 4 on 2 or more of the following PANSS items: delusions, conceptual disorganization, hallucinations, and unusual thought content at Baseline (Day 1).3. Subject must have a CGI-S score ≥ 4 at Baseline (Day 1).
   3. Subject must not demonstrate a decrease (improvement) of ≥ 20% in the PANSS total score between Screening and Baseline visits, or the PANSS total score falls below 80 at Baseline (Day 1).
   4. Subject must have a total score < 5 on the SAS at Baseline (Day 1).
   5. Subject must have a total score < 5 on the SAS at Baseline (Day 1).
   6. Subject must not answer "yes" to "Suicidal Ideation" Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) on the C-SSRS assessment at Baseline (ie, since last visit).
   7. Subject must meet all other inclusion and none of the exclusion criteria at Baseline (Day 1).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 245 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (6):
  - Woodland International Research Group, Little Rock, Arkansas
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - California Neuropsychopharmacology Clinical Research Institute-LA, LLC(CNRI- LA, LLC), Pico Rivera, California
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Pillar Clinical Research, LLC, Richardson, Texas
- Hungary (2):
  - Rehabilitacios Elmegyogyaszati osztaly, Gyöngyös
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
- Romania (4):
  - Bucharest
  - Centrul de Evaluare si Tratament al Toxicodependentelor pentru Tineri "Sfantul Stelian" - C.E.T.T.T. "Sf. Stelian", Bucharest
  - Spitalul Clinic de Neuropsihiatrie Craiova, Craiova
  - Institutul de Psihiatrie Socola Iasi, Sectia Clinica III Acuti, Sos. Bucium, Iași
- Russia (10):
  - State Budgetary Institution of Republic Karelia "Republican Psychiatric Hospital", Matrosy, Republic Karelia
  - Federal State Budgetary Scientific Instittuion "Scientific Center of Mental Health, Moscow
  - Saint Petersburg State Budgetary Institution of Healthcare "Psychiatric Hospital #1 named after P.P. Kashchenko", Saint Petersburg
  - City Psychiatric Hospital of St. Nikolay Chudotvorets, Saint Petersburg
  - FSBI Saint Petersburg Scientifc and Research Psychoneurological Instatitute named after V.M Bekhterev, Saint Petersburg
  - SPHI "City Mental Hospital #3 n.a. I.I.Skvortsov-Stepanov", Saint Petersburg
  - 300173524, Saint Petersburg
  - 300151369, Saratov
  - SBEI HPE "Smolensk State Medical University" of the MoH of the RF, Smolensk
  - 300195230, Yekaterinburg
- Ukraine (11):
  - Ch of Psychiatry, Narcology and Med Psychol, Ivano-Frankivsk
  - Dept of Crisis Cond & Primary Psych Episode #1, Ivano-Frankivsk
  - Psychiatric Department of Primary Psychotic Episodes, Kharkiv
  - Unit of Emergency Psychiatry and Narcology, Kharkiv
  - Dept of Psychiarty #3 (male) and #10 (female), Kherson
  - TMA Psychiatry in Kyiv Center of NT & Rehabilitation of Psychotic Conditions, Kyiv
  - CI Odesa Regional Medical Center of Mental Health, Odesa
  - Femal Dept #11, Male Dept #12, Smila
  - Ch of Neurology, Psychiatry, Narcology and MP, Ternopil
  - Dept of Psychiatry, Uzhhorod
  - Ch of Psychiatry and Narcology, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com

REFERENCES:
- [Derived] Halff EF, Rutigliano G, Garcia-Hidalgo A, Howes OD. Trace amine-associated receptor 1 (TAAR1) agonism as a new treatment strategy for schizophrenia and related disorders. Trends Neurosci. 2023 Jan;46(1):60-74. doi: 10.1016/j.tins.2022.10.010. Epub 2022 Nov 8. PMID 36369028
- [Derived] Koblan KS, Kent J, Hopkins SC, Krystal JH, Cheng H, Goldman R, Loebel A. A Non-D2-Receptor-Binding Drug for the Treatment of Schizophrenia. N Engl J Med. 2020 Apr 16;382(16):1497-1506. doi: 10.1056/NEJMoa1911772. PMID 32294346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | SEP-363856
Started | 125 | 120
Subjects Continued Into Extension Study | 79 | 78
Completed | 99 | 94
Not Completed | 26 | 26
Not completed — Adverse Event | 8 | 10
Not completed — Lack of Efficacy | 4 | 5
Not completed — Death | 0 | 1
Not completed — PROTOCOL DEVIATION | 0 | 1
Not completed — Withdrawal by Subject | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SEP-363856 | Total
Number analyzed (Participants) | 125 | 120 | 245
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 123 | 120 | 243
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.6 (6.07) | 30.0 (5.76) | 30.3 (5.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 89
  Male | 79 | 77 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 119 | 115 | 234
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 20 | 19 | 39
  White | 104 | 96 | 200
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  >=18 - <25 years | 29 | 26 | 55
  >=25 - <=40 years | 96 | 94 | 190
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] | 172.7 (7.78) | 173.0 (8.50) | 172.8 (8.12)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] | 73.74 (12.645) | 75.23 (15.768) | 74.47 (14.250)
Baseline Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 24.71 (3.727) | 25.01 (4.238) | 24.86 (3.981)
Baseline Body Mass Index (BMI) Group [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 1 | 4 | 5
  >=18.5 - <25.0 kg/m^2 | 70 | 59 | 129
  >=25.0 - <30.0 kg/m^2 | 43 | 41 | 84
  >=30.0 kg/m^2 | 11 | 16 | 27
Baseline Waist Circumference (cm) [Mean (Standard Deviation); unit: cm] | 84.18 (12.186) | 85.21 (14.191) | 84.68 (13.189)
Country [Count of Participants; unit: Participants]
  Hungary | 6 | 6 | 12
  Romania | 5 | 5 | 10
  Russia | 52 | 46 | 98
  Ukraine | 37 | 36 | 73
  United States | 25 | 27 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 4
Description: PANSS comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -9.7 (1.61) | -17.2 (1.66)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Net) = -7.5, 95% CI 2-sided [-11.9 to -3.0], Standard Error of Mean 2.23

2. Secondary Outcome: Change From Baseline in Clinical Global Impression - Severity (CGI-S) Score at Week 4
Description: The CGI-S a single-item clinician-rated assessment of the subject's current illness state on a 7-point scale (score range: 1-7), where a higher score is associated with greater illness severity.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -0.5 (0.09) | -1.0 (0.09)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.5, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.12

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Subscale Score at Week 4
Description: PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS Positive subscale score means more severe outcome.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -3.9 (0.51) | -5.5 (0.53)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p = 0.019, Mixed Models Analysis; Mean Difference (Net) = -1.7, 95% CI 2-sided [-3.1 to -0.3], Standard Error of Mean 0.71

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Subscale Score at Week 4
Description: PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS Negative subscale score means more severe outcome.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -1.6 (0.41) | -3.1 (0.42)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p = 0.008, Mixed Models Analysis; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.6 to -0.4], Standard Error of Mean 0.55

5. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) General Psychopathology Subscale Score at Week 4
Description: PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS General Psychopathology subscale score means more severe outcome.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -4.7 (0.84) | -9.0 (0.87)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -4.3, 95% CI 2-sided [-6.6 to -2.0], Standard Error of Mean 1.15

6. Secondary Outcome: Change From Baseline in Brief Negative Symptom Scale (BNSS) Total Score at Week 4
Description: The BNSS is a rating scale to measure the current level of severity of negative symptoms in schizophrenia and schizoaffective disorder. The measure is comprised of 13 individual items organized in 6 subscales. The 13 individual items provide a composite total score (ranging from 0 to 78). Each of the items are scored on a Likert-type 7-point scale from 0 - 6, where values of 0 indicates symptom is absent and a value of 6 means the symptom is a severe form. Higher BNSS total score means more severe outcome.
Time Frame: Baseline, Week 4
Population: Subjects who had BNSS total score data available are included in this analysis.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 119 | 113
Units on a scale | -2.7 (0.91) | -7.1 (0.95)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -4.3, 95% CI 2-sided [-6.8 to -1.8], Standard Error of Mean 1.26

7. Secondary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 4
Description: The MADRS is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts. Each item is scored in a range of 0 to 6 points, with higher scores indicating increased depressive symptoms. Total score will be equal to the sum of the 10 items (range between 0 and 60). Higher MADRS total score means more severe outcome.
Time Frame: Baseline, Week 4
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Units on a scale | -1.6 (0.57) | -3.3 (0.59)
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p = 0.020, Mixed Models Analysis; Mean Difference (Net) = -1.8, 95% CI 2-sided [-3.2 to -0.3], Standard Error of Mean 0.75

8. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS) Response at Week 4, Defined as a 20% or Greater Improvement From Baseline in PANSS Total Score
Description: PANSS is comprised of 30 items and 3 subscales (Positive, Negative, General Psychopathology). An anchored Likert scale from 1 - 7, where values of 2 and above indicate the presence of progressively more severe symptoms, is used to score each item. Individual items are then summed to determine scores for the 3 subscales, as well as a total score. PANSS Positive subscale score range: 7-49. PANSS Negative subscale score range: 7-49. PANSS General Psychopathology subscale score range: 16-112. PANSS total score range: 30-210. Higher PANSS total score means more severe outcome.
Time Frame: Baseline, Week 4
Population: Subjects who had PANSS total score data available at both Baseline and Week 4 are included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 100 | 96
Participants | 44 | 62
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio (OR) = 2.645, 95% CI 2-sided [1.422 to 4.921]

9. Secondary Outcome: The Incidence of Overall AEs, Serious AEs (SAEs) and AEs (or SAEs) Leading to Discontinuation
Time Frame: From first dose of study drug to last study visit, up to 5 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Participants
  Overall Adverse Events (AEs) | 63 | 55
  Serious Adverse Events (SAEs) | 3 | 2
  AEs/SAEs leading to discontinuation from study | 8 | 11
  AEs/SAEs leading to discontinuation of study drug | 8 | 10

10. Secondary Outcome: Frequency of Subjects With Suicidal Ideation Using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS is a tool designed to systematically assess and track suicidal behavior and suicidal ideation for life time, one month prior to the screening visit for suicidal ideation and 6 months prior to the screening visit for suicidal behavior, and throughout the study. The strength of this suicide classification system is in its ability to comprehensively identify suicidal events while limiting the over-identification of suicidal behavior.
Time Frame: Overall post-Baseline double-blind treatment period, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Participants | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Other; p = 0.498, Fisher Exact

11. Secondary Outcome: Frequency of Subjects With Suicidal Behavior Using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: as for outcome 10
Time Frame: Overall post-Baseline double-blind treatment period, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Participants | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Other; p > 0.999, Fisher Exact

12. Secondary Outcome: Frequency of Subjects With Suicidality Using the Columbia - Suicide Severity Rating Scale (C-SSRS)
Description: as for outcome 10
Time Frame: Overall post-Baseline double-blind treatment period, up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | SEP-363856
Number analyzed (Participants) | 125 | 120
Participants | 2 | 0
Statistical Analysis 1: Comparison: Placebo vs SEP-363856; Test type: Other; p = 0.498, Fisher Exact

ADVERSE EVENTS:
Time Frame: 5 weeks (from first dose of study drug to last study visit)
Arm/Group | Placebo | SEP-363856
All-Cause Mortality (participants affected / at risk) | 0/125 | 1/120
Serious Adverse Events (participants affected / at risk) | 3/125 | 2/120
Other Adverse Events (participants affected / at risk) | 47/125 | 35/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | SEP-363856 (N=120)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1)
Schizophrenia (Psychiatric disorders) | 3 (3) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=125) | SEP-363856 (N=120)
Headache (Nervous system disorders) | 15 (18) | 11 (15)
Somnolence (Nervous system disorders) | 6 (6) | 8 (8)
Anxiety (Psychiatric disorders) | 9 (12) | 2 (2)
Insomnia (Psychiatric disorders) | 13 (20) | 4 (5)
Schizophrenia (Psychiatric disorders) | 7 (8) | 7 (7)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (7)
Agitation (Psychiatric disorders) | 6 (6) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/82/NCT02969382/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-28): https://cdn.clinicaltrials.gov/large-docs/82/NCT02969382/SAP_001.pdf